CLINICAL TRIAL: NCT06356610
Title: A Randomized, Controlled, Six-way Crossover Clinical Study To Characterize The Nicotine Pharmacokinetics And Subjective Effects Of Four Heated Tobacco Products In Adult Menthol And Nonmenthol Cigarette Smokers
Brief Title: Pharmacokinetic and Subjective Effects of Heated Tobacco Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ALCS-REG-23-08-HT
Record Dates: First submitted 2024-03-12; First posted 2024-04-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2024-10

CONDITIONS: Tobacco Use
Keywords: Tobacco; Smoking; Heated tobacco
MeSH Terms: conditions — Tobacco Use; Smoking | interventions — Nicotine Chewing Gum; Menthol

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, six-way crossover clinical study to characterize the nicotine PK and subjective effects of HTPs (2 menthol varieties, Products A and B; 2 tobacco flavor varieties, Products C and D). The study will include participants' UBCC (Product F) and a nicotine gum (Product E) as high and low abuse liability reference products. Sponsor will prepare the randomization schedule. On Day -1 participants will be randomized at 1:1:1:1:1:1 ratio into 1 of 6 sequences as listed below. At least 60 participants will be randomized to ensure approximately 48 completed participants, with approximately 24 menthol and 24 non-menthol cigarette smokers. Participants will be stratified by sex and cigarette type for each of the sequences. A 6x6 Latin Square with the following sequences will be used for the randomization: Sequence 1 = ABFCED Sequence 2 = BCADFE Sequence 3 = CDBEAF Sequence 4 = DECFBA Sequence 5 = EFDACB Sequence 6 = FAEBDC.
Who Masked: Participant
Masking Description: Study participants will know when they are using their UBCC (usual brand combustible cigarette) and the nicotine gum. However, participants will not be informed of which Ploom® HTS (heated tobacco stick) product they are using. Participants will not see the stick or device packaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Randomization Sequence 1: ABFCED (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product A Test Product B Reference Product F Test Product C Reference Product E Test Product D
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Reference Product E; Other: Reference Product F
- Randomization Sequence 2: BCADFE (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product B Test Product C Test Product A Test Product D Reference Product F Reference Product E
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Reference Product E; Other: Reference Product F
- Randomization Sequence 3: CDBEAF (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product C Test Product D Test Product B Reference Product E Test Product A Reference Product F
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Reference Product E; Other: Reference Product F
- Randomization Sequence 4: DECFBA (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Test Product D Reference Product E Test Product C Reference Product F Test Product B Test Product A
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Reference Product E; Other: Reference Product F
- Randomization Sequence 5: EFDACB (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Reference Product E Reference Product F Test Product D Test Product A Test Product C Test Product B
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Reference Product E; Other: Reference Product F
- Randomization Sequence 6: FAEBDC (Experimental): Usage of Test and Reference study products in controlled use and ad libitum use sessions during the 6 day in-clinic period in following order:
  Reference Product F Test Product A Reference Product E Test Product B Test Product D Test Product C
  Interventions: Other: Test Product A; Other: Test Product B; Other: Test Product C; Other: Test Product D; Other: Reference Product E; Other: Reference Product F

INTERVENTIONS:
Other: Test Product A — Use of Test Product A in controlled use and ad libitum use sessions
  Other Names: Ploom® 3.1 HTP - Menthol HTS; MX3 (681)
Other: Test Product B — Use of Test Product B in controlled use and ad libitum use sessions
  Other Names: Ploom® 3.1 HTP - Menthol HTS; MX5 (706)
Other: Test Product C — Use of Test Product C in controlled use and ad libitum use sessions
  Other Names: Ploom® 3.1 HTP - Tobacco HTS; R8 (120)
Other: Test Product D — Use of Test Product D in controlled use and ad libitum use sessions
  Other Names: Ploom® 3.1 HTP - Tobacco HTS; RX4 (953)
Other: Reference Product E — Use of Reference Product E in controlled use and ad libitum use sessions
  Other Names: Nicorette® 4 mg Mint Nicotine Gum
Other: Reference Product F — Use of Reference Product F in controlled use and ad libitum use sessions
  Other Names: Combustible Cigarette (menthol or nonmenthol), participant's usual brand

SUMMARY:
This is a randomized, controlled, six-way crossover clinical study to characterize the nicotine PK (pharmacokinetic) and subjective effects of HTPs (Heated Tobacco Products) comprised of 2 menthol varieties and 2 tobacco flavor varieties (Ploom® HTPs, Japan Tobacco Inc.) in adult menthol and non-menthol combustible cigarette smokers (males and females between the ages of 22 and 65). The study will include participants' UBCC (Usual Brand Combustible Cigarette) and a nicotine gum (Nicorette®) as high and low abuse liability reference products, respectively, to the HTP. Study participation is expected to last up to 34 days, including a 28-day screening period (that includes a 5-day at-home HTP product trial period), and a 6-day in-clinic confinement period (from Check-in [Day -1] through the end-of-study [EOS] visit on Day 6).

DETAILED DESCRIPTION:
This is a randomized, controlled, six-way crossover clinical study to characterize the nicotine PK and subjective effects of HTPs (2 menthol varieties, Products A and B; 2 tobacco flavor varieties, Products C and D) in adult menthol and non-menthol combustible cigarette smokers. The study will include participants' UBCC (Product F) and a nicotine gum (Product E) as high and low abuse liability reference products, respectively, to the HTP. The study will include generally healthy adult males and females who smoke factory manufactured combustible cigarettes. This study will recruit approximately 60 participants (composed of approximately 30 menthol and 30 non-menthol adult smokers) in an attempt to obtain approximately 48 study completed participants (approximately 24 menthol and 24 non-menthol smokers). Adult participants will be between 22 and 65 years of age at screening, inclusive. Participants must have a history of smoking ≥ 10 to ≤ 30 menthol or non-menthol cigarettes daily for at least 12 months prior to screening.

Enrolled participants will be randomized based on sex and their UBCC (menthol or non-menthol) to one of 6 product use sequences.

Screening will occur within 28 days prior to Day 1 and includes administering the FTCD (Fagerstrom Test for Cigarette Dependence), standard safety procedures, collection of baseline information, and a 5-day at-home HTP product trial period.

Enrollment visit (Day -6) will occur 5 days prior to Check-in (Day -1). Participants will receive the Ploom® HTP products for at-home product acclimation to become familiar with the product during the next 5 days. Training on how to use the Ploom® HTP device will be provided to each participant at the Enrollment visit. Participants will receive all four varieties of HTS on Day -6 and begin the at-home product trial. Participants are required to use each HTS variety at least once a day ad libitum for a minimum of 20 HTS uses over 5 days.

Participants will check-in on the morning of Day -1. Product use sequence randomization and assignment will also occur on Day -1. Participants will be randomized based on sex and their UBCC (menthol or non-menthol) to one of six product use sequences. Once participants are randomized to a product use sequence, product use sessions in confinement will start. Participants will remain in confinement at the clinic until completion of all study activities on Day 6.

Starting on Day -1 (following Check-in) through Day 5, depending on the randomized product use sequence, participants will use their assigned product (HTP, UBCC, or nicotine gum) during an afternoon product use session. Participants will use the same assigned product to be tested during the next day's morning ad libitum product use PK test session (e.g., if a participant is assigned to Product A [HTP] as the product to be used in the morning ad libitum product use PK test session on Day 1, the participant will use Product A [HTP] during the afternoon product use session on Day -1). The afternoon product use session should be no more than approximately 6 hours long. Participants will be required to use the assigned study product at least once, but no more than six HTS, UBCC, or nicotine gum ad libitum per daily afternoon product use sessions. Participants will then be required to abstain from any tobacco- or nicotine-containing products for at least 12 hours prior to the start of the following morning's ad libitum product use PK test session. Morning ad libitum product use PK test sessions will occur on the mornings of Days 1, 2, 3, 4, 5, and 6 (for a total of 6 morning ad libitum product use PK test sessions).

During the morning ad libitum product use PK test session, participants will use the assigned study product per their assigned product use sequence. Participants will use a single UBCC or HTP for 5 minutes ad libitum or use the nicotine gum for 30 minutes per product use instruction. Blood samples for PK will be collected prior to and for 3 hours following the start of each morning ad libitum product use PK test session. Heart rate measurements will be taken at specified time points during each morning ad libitum product use PK test session. In addition, participants will complete subjective effects questionnaires (Product Liking, Tobacco/Nicotine Withdrawal, Direct Effects of Product, Use Product Again, and mCEQ) at designated time points during each morning ad libitum product use PK test session. Participants will remain in confinement starting with Check-in on Day -1 until discharge after all study activities are completed on Day 6. Participants will not be forced to use the tobacco/nicotine products at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be informed of the nature and risks of the study and voluntarily give written informed consent prior to screening.
2. Healthy adult males and females ≥ 22 and ≤ 65 years of age, inclusive, at screening.
3. Participants must self-report currently smoking menthol or non-menthol factory manufactured combustible cigarettes. Participants will have a history of smoking ≥ 10 to

   ≤ 30 menthol or non-menthol factory manufactured combustible cigarettes daily for at least 12 months prior to screening. Prior to screening, brief periods (i.e., up to 7 consecutive days) of non-smoking within 90 days before Check-in (e.g., due to illness or participation in a clinical study where tobacco use was prohibited) will not be exclusionary at the discretion of the Investigator (other non-daily tobacco use, except for heated tobacco use, within 30 days prior to screening are not exclusionary).
4. Participants must be generally healthy, free of lifetime malignant tumors, and without clinically significant abnormalities as assessed by the Investigator based on the review of medical and surgical history, physical examination, vital signs, 12-lead ECG, and laboratory evaluations conducted at screening and Check-in, as applicable (refer to Table 1). A single repeat measurement/test may be performed to confirm vital signs, 12-lead ECG, and clinical laboratory tests abnormalities (i.e., to confirm that a participant is eligible).
5. Screening and Check-in systolic/diastolic blood pressure ≤ 150/90 mmHg measured after being seated quietly for at least 10 minutes. Two rechecks may be performed at the Investigator's discretion.
6. Urine cotinine ≥ 500 ng/mL at screening.
7. Exhaled carbon monoxide ≥ 10 ppm at screening.
8. Negative pregnancy test at screening and Check-in (Day -1) for all female participants.
9. Female participants who are sexually active and of childbearing potential (i.e., not surgically sterile at least 6 months prior to Check-in nor post-menopausal with amenorrhea for at least 1 year prior to Check-in and FSH levels consistent with postmenopausal status) must not be lactating and must have been using one of the following forms of contraception from 3 months before first study product administration through 30 days after the final administration of study product:

   * hormonal (e.g., oral, vaginal ring, transdermal patch, implant, injection) consistently for at least 3 months prior to Check-in, when used in combination with male condoms with spermicide (use of NuvaRing® is at the Investigator's discretion)
   * double barrier (e.g., condom with spermicide or diaphragm with spermicide) consistently for at least 2 weeks prior to Check-in
   * intrauterine device or system (utilize Investigator discretion regarding use of hormonal or nonhormonal devices) for at least 3 months prior to Check-in
   * exclusive partner who is clinically sterile (i.e., documented infertility or surgical sterilization; see below for additional information on sterility) or has been vasectomized for at least 6 months (inclusive) prior to Check-in Note: Sexual abstinence, defined as refraining from intercourse, is allowed when this is in line with the preferred and usual lifestyle of the participant. Female participants of childbearing potential who are not currently engaging in heterosexual intercourse must agree to use one of the above methods of birth control through completion of study, in the event that they have heterosexual intercourse during the course of the study.
10. Female participants who are of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to Check-in:

    * hysteroscopic sterilization with documentation of success with hysterosalpingogram
    * bilateral tubal ligation or bilateral salpingectomy
    * hysterectomy
    * bilateral oophorectomy
    * Essure® or be post-menopausal with amenorrhea for at least 1 year prior to Check-in and confirmed by FSH levels consistent with post-menopausal status.
11. Able to communicate effectively with the study personnel and willing to comply with the requirements of the study.
12. Willing and able to use all of the study products. This includes product use during the at-home product trial and the in-confinement product use sessions. If participants are unwilling to use or unable to tolerate any of the study products they will not participate in this study.

Exclusion Criteria:

1. Use of any HTPs within the past 30 days prior to the screening visit; occasional use (i.e., not daily use) of other types of tobacco- or nicotine-containing products other than factory manufactured combustible cigarettes (e.g., roll-your-own cigarettes, e-cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) are allowed within the past 30 days prior to screening.
2. Any postponement of a quit attempt to participate in the study; or any attempts to quit smoking in the 3 months prior to Day -1 (Check-in).
3. Self-reported puffers (i.e., smokers who draw smoke from the combustible cigarette into the mouth and throat but do not inhale).
4. Poor dentition that prevents participant from using nicotine gum.
5. History or presence of any type of malignant tumor or clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, pulmonary, immunologic, psychiatric, or cardiovascular disease, or any other condition that, in the opinion of the Investigator, would interfere with the absorption, distribution, metabolism, or excretion of cotinine or jeopardize the safety of the participant or impact the validity of the study results.
6. Current evidence or any history of congestive heart failure.
7. Any other condition or prior therapy that, in the Investigator's opinion, would make the participant unsuitable for the study, or unable or unwilling to comply with the study procedures.
8. Clinically significant abnormal vital sign, physical examination (including oral cavity an oropharynx), medical history, or clinical laboratory finding(s), in the opinion of the Investigator.
9. Positive test for human immunodeficiency virus (HIV)-1 or HIV-2; or hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) consistent with current infection at screening.
10. Diabetes mellitus that is not controlled by diet/exercise alone, in the opinion of the Investigator. Fasting plasma glucose > 126 mg/dL (7 mmol/L) is exclusionary. One recheck may be performed for fasting plasma glucose values > 126 mg/dL but < 200 mg/dL.
11. An acute illness (e.g., upper respiratory infection, viral infection) requiring treatment with prescribed medicines within 2 weeks prior to Check-in.
12. History of surgery or major trauma within 12 weeks of screening, or surgery planned during the study through EOS.
13. History of alcohol abuse or drug abuse within 24 months prior to Check-in.
14. Consumption of alcohol-containing food or beverages within 48 hours prior to Check-in.
15. Positive screen for alcohol (breath or urine) or any of the following drugs of abuse (urine), regardless of the reason of use: amphetamines, methamphetamines, opiates, cannabinoids, or cocaine at screening or Check-in.
16. Fever (i.e., body temperature > 100.5°F) at screening or Check-in; 1 recheck may be performed at the Investigator's discretion.
17. Body mass index (NHLBI) > 40.0 kg/m2 or < 18.0 kg/m2 at screening.
18. Estimated glomerular filtration rate < 80 mL/minute using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula (Medscape) at screening.
19. Serum alanine aminotransferase ≥ 1.5 times the upper limit of normal and/or aspartate aminotransferase ≥ 2.0 times the upper limit of normal at screening; 1 recheck may be performed at the Investigator's discretion.
20. Female participants who are pregnant (positive pregnancy test at screening or Check-in), lactating, or intend to become pregnant from screening through EOS.
21. Use of prescription or over-the-counter (OTC) bronchodilator medication (e.g., inhaled or oral β-agonists) for treatment of any illness within 12 months prior to Check-in.
22. Use of antibiotics within 2 weeks prior to Check-in. Also refer to Section 5.7.1.
23. Use of medications known or are suspected to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, buprenorphine, clofibrate, clotrimazole, desipramine, disulfiram, entacapone, fenofibrate, isoniazid, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine) within 14 days or 5 half-lives of the drug, whichever is longer, prior to Check-in.
24. Has taken other investigational drugs/products or participated in any clinical study for an investigational drug, device, biologic, or for a tobacco product within 30 days or 5 halflives (if known) of the investigational product's PK, pharmacodynamic, or biological activity (if known), whichever is longer, prior to first administration of study product in this study or is currently participating in another clinical study; or participation in > 2 ALCS-sponsored studies within the past 12 month period prior to Check-in.
25. Has received a vaccination within 14 days prior to Check-in.
26. Plasma donation within 7 days prior to Day 1.
27. Donation of ≥ 1 unit of blood or blood products (with the exception of plasma as noted), had significant blood loss > 450 mL, or received whole blood or a blood product transfusion within 56 days prior to Day -1.
28. Strenuous activity (as assessed by the Investigator) within 48 hours prior to Check-in.
29. Participant or a first-degree relative (i.e., parent, sibling, child, spouse) is a current or former employee of the tobacco industry or a named party or class representative in litigation with any tobacco company.
30. Participant or a first-degree relative (i.e., parent, sibling, child, spouse) is a current employee of the study site.
31. Unwilling or unlikely to comply with the requirements of the study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2024-02-06 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Plasma Nicotine Concentration Pharmacokinetic (PK) Measurement | Day 1 through Day 6
  Characterize PK parameters of nicotine in plasma during and after a single ad libitum use of HTP (two menthol and two tobacco flavor varieties) relative to UBCC and the nicotine gum. Plasma nicotine will be measured as ng/mL with baseline adjustment.
Product Liking of Heated Tobacco Products (HTP) | Day 1 through Day 6
  Characterize Product Liking of HTP (two menthol and two tobacco flavor varieties) during and after a single ad libitum use relative to UBCC and the nicotine gum by administering a Product Liking Questionnaire. This question is paired with a VAS (visual analog scale). The 100 mm VAS is anchored with 'Strongly Dislike' on the left, 'Neither Like nor Dislike' in the center and 'Strongly Like' on the right. Participants place a vertical line at a place along the VAS based on how he/she feels in the moment.
Tobacco Nicotine Withdrawal Questionnaire | Day 1 through Day 6
  Characterize subjective response to HTP (two menthol and two tobacco flavor varieties) during and after a single ad libitum use relative to UBCC and the nicotine gum through the administration of Tobacco Nicotine Withdrawal questionnaire adapted from Hughes and Hatsukami (1986). Each question will be paired with a 100 mm VAS. The VAS is anchored with "Not at All" on the left and "Extremely" on the right. Participants place a vertical line at a place along the VAS based on how he/she feels in the moment.
  Reference: Hughes JR, Hatsukami D (1986). Signs and symptoms of tobacco withdrawal. Archives of General Psychiatry. 43(3):289-94.
Direct Effects of Product Questionnaire | Day 1 through Day 6
  Direct Effects of Product Questionnaire contains items that were selected based on measures of product effects used in previous trials with conventional cigarettes and other tobacco products. Each question is paired with a 100 mm VAS. The VAS is anchored with "Not at ALL" on the left and "Extremely" on the right. Participants place a vertical line at a place along the VAS based on how he/she feels in the moment.
Use the Product Again Questionnaire | Day 1 through Day 6
  The Use the Product Again Questionnaire was adapted from abuse-deterrent drug formulation drug trials question "I would want to take this drug again." The question is paired with a 100 mm VAS. The VAS is anchored with "Definitely Would Not" on the left and "Definitely Would" on the right. Participants place a vertical line at a place along the VAS based on how he/she feels in the moment.
Modified Cigarette Evaluation Questionnaire (mCEQ) - Cigarette | Day 1 through Day 6
  The instructions for subjects are: Please mark the number that best represents how using the product made you feel (1 - not at all, 2 - very little, 3-a little, 4-moderately, 5-a lot, 6-quite a lot, 7-extremely)
Modified Cigarette Evaluation Questionnaire - HTP | Day 1 through Day 6
  Modified Cigarette Evaluation Questionnaire is further modified for heated tobacco product (mCEQ-HTP). The instructions to subjects for completion of the questionnaire are: Thinking about the study product that you used today, please mark the number that best represents how using the heated tobacco product made you feel (1- not at all, 2- very little, 3-a little, 4-moderately, 5-a lot, 6-quite a lot, 7-extremely).
Modified Cigarette Evaluation Questionnaire-NRT | Day 1 through Day 6
  Modified Cigarette Evaluation Questionnaire was further modified for oral tobacco derived nicotine products. The instructions for subjects are: Please mark the number that best represents how using the product made you feel (1-not at all, 2-very little, 3-a little, 4-moderately, 5-a lot, 6-quite a lot, 7-extremely).
Product Use for HTP-Units Dispensed | Day 1 through Day 6
  For the HTP use the number of units dispensed will be manually documented for the 5-minute ad libitum product use period during the morning ad libitum product use PK test session. During the afternoon product use session (6 hours max ad libitum product use) the number of units used will be manually documented for the 5-minute ad libitum product use.
Product Use for UBCC-Units Dispensed | Day 1 through Day 6
  For the UBCC use the number of units dispensed will be manually documented for the 5-minute ad libitum product use period during the morning ad libitum product use PK test session. During the afternoon product use session (6 hours max ad libitum product use) the number of units used will be manually documented for the 5-minute ad libitum product use.
Product Use for Nicotine Gum-Units Dispensed | Day 1 through Day 6
  For nicotine gum, the number of units dispensed will be manually documented for the 30-minute ad libitum product use during the morning ad libitum product use PK test session. During the afternoon product use sessions (6 hours max ad libitum product use), the number of units of nicotine gum dispensed will be documented manually.
Product Use for HTP-Puff Count | Day 1 through Day 6
  For HTP use the puff count will be the number of puffs per unit manually documented for the 5-minute ad libitum product use period during the morning ad libitum product use PK test session. During the afternoon product use session (6 hours max ad libitum product use) the puff count for each unit used will be manually documented for the 5-minute ad libitum product use.
Product Use for UBCC-Puff Count | Day 1 through Day 6
  For UBCC use the puff count measured as the number of puffs per unit will be manually documented for the 5-minute ad libitum product use period during the morning ad libitum product use PK test session. During the afternoon product use session (6 hours max ad libitum product use) the number of puffs per each unit used will be manually documented for the 5-minute ad libitum product use.
Physiological Heart Rate (HR) Assessment-HTP | Day 1 through Day 6
  Physiological HR assessments will be assessed at designated time points during the morning ad libitum HTP product use PK test sessions. The scheduled time points are to include -5, 5, 15, 30, 60 and 180 minutes during PK session. Heart rate measurements as beats per minute (BPM) will be performed prior to the blood draw (approximately 1 minute prior to the scheduled blood draw time point) when scheduled at the same time.
Physiological Heart Rate (HR) Assessment-UBCC | Day 1 through Day 6
  Physiological HR assessments will be assessed at designated time points during the morning ad libitum UBCC product use PK test sessions. The scheduled time points are to include -5, 5, 15, 30, 60 and 180 minutes during PK session. Heart rate measurements as beats per minute (BPM) will be performed prior to the blood draw (approximately 1 minute prior to the scheduled blood draw time point) when scheduled at the same time.
Physiological Heart Rate (HR) Assessment-Nicotine Gum | Day 1 through Day 6
  Physiological HR assessments will be assessed at designated time points during the morning ad libitum nicotine gum product use PK test sessions. The scheduled time points are to include -5, 5, 15, 30, 60 and 180 minutes during PK session. Heart rate measurements as beats per minute (BPM) will be performed prior to the blood draw (approximately 1 minute prior to the scheduled blood draw time point) when scheduled at the same time.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - QPS Bio-Kinetic, Springfield, Missouri
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No